CLINICAL TRIAL: NCT05179863
Title: Swiss Rare Disease Registry
Brief Title: Swiss Rare Disease Registry (SRDR)
Acronym: SRDR
Status: Recruiting | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: Federal Office of Public Health, Switzerland (Other Government); Universitäts-Kinderspital Zürich (Unknown); University Children's Hospital Basel (Other); Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Zürich (Other); Centre Hospitalier Universitaire Vaudois (Other); University Hospital, Geneva (Other); Proraris Allianz seltener Krankheiten (Unknown); Kosek National Coordination Rare Diseases Switzerland (Unknown); Orphanet Suisse (Unknown); University of Zurich (Other); Kantonsspital Aarau (Other); Ente Ospedaliero Cantonale, Bellinzona (Other); Cantonal Hospital of St. Gallen (Other); Ostschweizer Kinderspital (Other); University Hospital, Basel, Switzerland (Other); Balgrist University Hospital (Other); Centro Malattie Rare della Svizzera Italiana (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2017-02313
Record Dates: First submitted 2021-12-02; First posted 2022-01-05 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Rare Diseases
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 80 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient population: Children, adolescents, and adults with a high suspicion, or a confirmed diagnosis of a rare disease who are treated or living in Switzerland.

SUMMARY:
The SRDR is a national registry that records rare diseases in people of any age who live in Switzerland. It serves as a platform for scientists, health professionals, affected people, and politicians.The SRDR aims to collect epidemiological data on rare diseases, and data on changes to the diagnosis over time. The SRDR will further serve as a research platform and facilitate patient participation in national and international studies. The SRDR will promote harmonization of data and method between the numerous existing disease-specific registries in Switzerland, will strengthen the exchange with international rare disease registries for research and policy, and will build a network for communication for patients and health care providers.

DETAILED DESCRIPTION:
Background: In Europe a disease is considered rare when fewer than one in 2'000 people are affected. Today, more than 7'000 rare diseases are known. Although scarce, rare diseases all together affect approximately 5-8% of the people around the world. In Switzerland, more than 500'000 people live with a rare disease. Clinical and epidemiological studies on rare diseases in Switzerland are lacking. Little is known about diagnostics, efficient treatment, and the course of rare diseases.

The cantonal Ethics Committee of Bern approved the SRDR project (project ID: 2017-02313, observational study, risk category A).

Objectives: The overall goal of the SRDR is to improve the care situation of people living with a rare disease in Switzerland. The development of a national registry to collect representative and complete data from children and adults with a rare disease in Switzerland helps to achieve this overall goal.

Primary objectives of the SRDR project:

1. Collect epidemiological data on rare diseases from all patients with rare diseases in Switzerland (incidence, prevalence, survival, mortality).
2. Collect data on quality of health care and outcomes (diagnosis, management, outcomes, quality indicators, treating institutions).
3. Setup a research platform for clinical, epidemiological, basic, and translational research on all rare diseases.
4. Facilitate patients to participate in national and international studies.
5. Promote harmonisation of data and methods between the numerous existing disease-specific registries in Switzerland.
6. Strengthen exchange with international rare disease registries for research and policy.
7. Build a network for communication, for patients and health care providers.

Procedure: After a person has been diagnosed with a rare disease, the medical staff inform the patient and/or the legal representative orally about the SRDR and its purpose during regular consultation. The medical staff will hand over the written age-appropriate patient information and the informed consent form. Patient organizations and the staff from the SRDR also have the possibility to inform people about the SRDR. Further, patients have the possibility to use a secure web-based application for self-notification.

The patient or/and the legal representative have 6 weeks to give or refuse the informed consent. Patients who wish to participate sign the consent form and are then registered in the SRDR. If a patient or/and legal representative do neither refuse registration nor sign informed consent within 6 weeks, the data will be registered. If a patient does not wish to participate, only a minimal anonymous data set is recorded.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a rare disease
* High suspicion of a rare disease
* Treated or living in Switzerland
* Signed informed consent

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals with a high suspicion, or a confirmed diagnosis of a rare disease who are treated or living in Switzerland.
Sampling Method: Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2071-01 (Estimated); Study Completion 2071-01 (Estimated)

PRIMARY OUTCOMES:
Personal Data | At diagnosis (age 0-99 years)
  Registering patients personal data
Diagnosis | At diagnosis (age 0-99 years)
  Orpha Code of the diagnosed rare disease
Date of Diagnosis | At diagnosis (age 0-99 years)
  Date on which the diagnosis was made
Disease History | At registration (age 0-99 years)
  History of first occurrence of symptoms
Diagnostic Method | At diagnosis (age 0-99 years)
  Diagnostic method that was decisive for the diagnosis
Molecular genetic information | At diagnosis (age 0-99 years)
  Name of affected genes and mutations
Other Registries | At registration (age 0-99 years)
  Name of other national or international registries the patient is registered

CONTACTS AND LOCATIONS:
Overall Officials: Claudia E Kuehni, Prof. MD, Principal Investigator — Institute of Social and Preventive Medicine (ISPM)
Locations (20):
- Switzerland (20):
  - Kantonsspital Aarau, Pädiatrie, Aarau
  - Kantonsspital Aarau, Aarau
  - Center for Rare Diseases, Basel, Basel
  - Universitäs-Kinderspital beider Basel, UKBB, Basel
  - Universitätsspital Basel, USB, Basel
  - Centro Malattie Rare della Svizzera Italiana, Bellinzona
  - Center for Rare Diseases, Inselspital, Bern
  - University of Bern, Inselspital Bern, Bern
  - Center for Rare Diseases, Geneva, Geneva
  - Hôpitaux universitaires de Genève, HUG, Geneva
  - Center for Rare Diseases, Lausanne, Lausanne
  - Centre hospitalier universitaire vaudois, CHUV, Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Ostschweizer Kinderspital, Sankt Gallen
  - Ostschweizer Zentrum für seltene Krankheiten, Pädiatrie, Sankt Gallen
  - Ostschweizer Zentrum für seltene Krankheiten, Sankt Gallen
  - Center for Rare Diseases, Zurich, Zurich
  - Universitäts-Kinderspital Zürich, Kispi, Zurich
  - Universitätsklinik Balgrist, Zurich
  - Universitätsspital Zürich, USZ, Zurich